CLINICAL TRIAL: NCT02147301
Title: Prospective Phase II Study of Chemoembolization With Doxorubicin-Eluting Microspheres for Liver Transplantation Candidates With Hepatocellular Carcinoma and Marginal Hepatic Reserve
Brief Title: TACE Using Doxorubicin-eluting Beads for Patients With HCC and Marginal Hepatic Reserve
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Risk to benefit ratio is not acceptable
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Nicholas Fidelman, MD, Principal Investigator, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 124520
Record Dates: First submitted 2014-05-19; First posted 2014-05-26 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Hepatocellular Carcinoma; Chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DEB-TACE (Experimental): Doxorubicin Eluting Bead Transarterial Chemoembolization (DEB-TACE):
  Doxorubicin-loaded LC Beads® are administered via a co-axially placed commercially available hepatic artery catheter into hepatic arteries targeted for treatment. Procedure is performed under direct fluoroscopic visualization until stasis of arterial flow is achieved or until a total of 4 ml of microspheres have been administered, whichever occurs first
  Interventions: Device: LC Bead

INTERVENTIONS:
Device: LC Bead — Doxorubicin Eluting Bead Transarterial Chemoembolization (DEB-TACE):
  Doxorubicin-loaded LC Beads® are administered via a co-axially placed commercially available hepatic artery catheter into hepatic arteries targeted for treatment. Procedure is performed under direct fluoroscopic visualization until stasis of arterial flow is achieved or until a total of 4 ml of microspheres have been administered, whichever occurs first.
  Other Names: DC Bead

SUMMARY:
TACE is frequently offered to patients with baseline hepatic dysfunction with the purpose of diminishing hepatic tumor burden while patients await transplantation. Without this therapeutic measure, disease may progress beyond UNOS T2 criteria required for organ allocation.

The purpose of the study is to determine whether transarterial chemoembolization using doxorubicin-eluting beads (DEB-TACE) can be used safely and effectively to treat patients with liver-only hepatocellular carcinoma (HCC) and baseline hepatic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female patients, age 18 years of age or older
2. Diagnosis of liver-only HCC based on European Association for the Study of the Liver (EASL) criteria (radiographic lesion appearance on contrast-enhanced CT or MRI, i.e. enhancement on early arterial phase, washout on portal venous phase with or without associated elevation of serum alpha-fetoprotein (AFP) level >200 Units Per Millilitre (U/ml)) or histologic confirmation of HCC diagnosis, whichever is applicable.
3. UNOS stage T1, T2, or T3 disease.
4. Candidates for liver transplantation (listed or screened) according to one of the following criteria:

   1. Milan criteria (one lesion < 5cm or 3 or fewer lesions each < 3cm),
   2. UCSF Downstaging criteria (one lesion less than 8 cm or 2-3 lesions each less than 5 cm with sum of maximum dimensions less than 8 cm, or 4-5 lesions each less than 3 cm with sum of maximum dimensions less than 8 cm)
   3. University of California, San Francisco (UCSF) All-Comers criteria (UNOS stage T3 disease beyond UCSF Downstaging Criteria).
5. At least one measurable site of disease in the liver according to RECIST version 1.1 and odified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria.
6. At least one of the following clinical, laboratory, or imaging parameters:

   1. Mild or moderate ascites
   2. Serum bilirubin ≥ 3 mg/dl but less than 6 mg/dl
   3. Aspartate aminotransferase (AST) > 5 times upper limit of normal (ULN) but < 10 times ULN
   4. Alanine aminotransferase (ALT) > 5 times upper limit of normal (ULN) but < 10 times ULN
   5. International normalized ratio for prothrombin time (INR) >1.5 but ≤ 2.5
   6. Portal vein thrombosis (branch or main)
   7. Functioning transjugular intrahepatic portosystemic shunt (TIPS) or surgical portosystemic shunt
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.

Exclusion Criteria:

1. Liver-directed therapy (chemoembolization, radioembolization, bland embolization, ablative therapy) within 4 weeks of DEB-TACE.
2. Previous liver transplantation.
3. Serum bilirubin ≥ 6 mg/dl
4. AST > 10 times upper normal limit
5. ALT > 10 times upper normal limit
6. INR > 2.5
7. Serum creatinine > 1.5 mg/dl
8. Macrovascular tumor invasion of portal and/or hepatic vein(s)
9. Extracapsular tumor extension
10. Extrahepatic disease
11. Hepatic encephalopathy refractory to medical therapy
12. Active uncontrolled infection
13. Imaging evidence of common bile duct obstruction
14. Previous sphincterotomy or bilio-enteric anastomosis
15. Significant hepatic arterial to portal vein shunting in the area to be treated.
16. Symptomatic congestive heart failure (CHF)
17. Allergy to or intolerance of prior doxorubicin-based TACE
18. Allergy to or intolerance to iodinated contrast media despite standard of care pre-medication
19. Any contraindications to treatment with LC Bead™ device (e.g. patients with large diameter arteriovenous shunts or patients with a right-to-left shunt).
20. Systemic therapy with sorafenib or other systemic chemotherapeutic agent(s) less than 1 week prior to first planned DEB-TACE.
21. Active second malignancy other than non-melanoma skin cancer or cervical carcinoma in situ. (Patients with history of malignancy are not considered to have a "currently active" malignancy if they have completed therapy and are now considered by their physician to be at less than 30% risk for relapse.)
22. Uncontrolled intercurrent illness including, but not limited to: Ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, uncontrolled peripheral vascular disease, myocardial infarction within preceding 12 months, cerebrovascular accident within preceding 12 months, pulmonary disease impairing functional status or requiring oxygen, impairment in gastrointestinal function that may affect or alter absorption of oral medications (such as malabsorption or history of gastrectomy or bowel resection).
23. Pregnant or lactating women are excluded from this study because of the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with DEB-TACE, breastfeeding must be discontinued for eligibility.
24. Psychiatric illness, other significant medical illness, or social situation which, in the investigator's opinion, would limit compliance or ability to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Fidelman, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 patients were enrolled and completed study.
Period: Overall Study
Arm/Group | DEB-TACE
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- DEB-TACE #1: Doxorubicin Eluting Bead Transarterial Chemoembolization (DEB-TACE):
  Doxorubicin-loaded LC Beads® are administered via a co-axially placed commercially available hepatic artery catheter into hepatic arteries targeted for treatment. Procedure is performed under direct fluoroscopic visualization until stasis of arterial flow is achieved or until a total of 4 ml of microspheres have been administered, whichever occurs first
  1st debtace treatment
Arm/Group | DEB-TACE #1
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Best Observed Radiographic Response Rate (Measured by mRECIST)
Description: Best observed radiographic response rate to Doxorubicin Eluting Bead Transarterial Chemoembolization (DEB-TACE) by modified Response Evaluation Criteria in Solid Tumors (mRECIST) was defined as number of patients who had CR, PR, or SD as their best observed response divided by total number of patients with at least one available CT or MRI. Definition of mRECIST for Hepatocellular Carcinoma (HCC). Complete response (CR) = Disappearance of any intratumoral arterial enhancement in all target lesions. Partial response (PR)=At least a 30% decrease in sum of diameters of viable (enhancement in arterial phase) target lesions, taking as reference baseline sum of diameters of target lesions. Stable disease (SD)=Any cases that do not qualify for either partial response or progressive disease. Progressive disease (PD)=An increase of at least 20% in the sum of the diameters of viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enh
Time Frame: 1 year
Population: Best observed radiographic response for all patients who had at least one follow-up cross-sectional imaging study
Measure: Count of Participants; unit: Participants
Groups:
- DEB-TACE: Doxorubicin Eluting Bead Transarterial Chemoembolization (DEB-TACE):
  Doxorubicin-loaded LC Beads® are administered via a co-axially placed commercially available hepatic artery catheter into hepatic arteries targeted for treatment. Procedure is performed under direct fluoroscopic visualization until stasis of arterial flow is achieved or until a total of 4 ml of microspheres have been administered, whichever occurs first
  LC Bead: Doxorubicin Eluting Bead Transarterial Chemoembolization (DEB-TACE):
  Doxorubicin-loaded LC Beads® are administered via a co-axially placed commercially available hepatic artery catheter into hepatic arteries targeted for treatment. Procedure is performed under direct fluoroscopic visualization until stasis of arterial flow is achieved or until a total of 4 ml of microspheres have been administered, whichever occurs first.
Arm/Group | DEB-TACE
Number analyzed (Participants) | 16
Participants
  Complete response | 4
  Partial response | 6
  Stable disease | 4
  Progressive disease | 2

2. Primary Outcome: Number of Patients Who Developed New Severe Adverse Events
Description: Number of patients who developed new severe adverse events according to NCI CTCAE version 4.0
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | DEB-TACE
Number analyzed (Participants) | 17
participants
  Ascites | 1
  Edema of limbs | 2
  Hepatic failure | 4
  Pain | 2
  Hyperbilirubinemia | 3
  AST elevation | 3
  Hyponatremia | 4
  Anemia | 2
  Thrombocytopenia | 3
  Creatinine elevation | 1

3. Secondary Outcome: Best Observed Objective Radiographic Response by mRECIST
Description: Best observed objective radiographic response was defined as the number of patients who had a complete response or partial response divided by total number of evaluable patients.
  Measured by mRECIST (see mRECIST definition in the description of the primary objective).
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | DEB-TACE
Number analyzed (Participants) | 16
participants | 10

4. Secondary Outcome: Time to Untreatable Progression (TTUP)
Description: TTUP is defined as time (months) from the first on-study DEB-TACE to development of radiographic disease progression untreatable by liver-directed percutaneous or surgical methods (by mRECIST).
Time Frame: 1 year
Population: months
Measure: Median (Full Range); unit: Months
Arm/Group | DEB-TACE
Number analyzed (Participants) | 17
Months | 9.7 [1.4 to 30.4]

5. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression was defined as the period of time from the first on-study DEB-TACE to radiographic disease progression at any site by mRECIST.
Time Frame: 1 year
Measure: Median (Full Range); unit: Months
Arm/Group | DEB-TACE
Number analyzed (Participants) | 17
Months | 5.6 [0.9 to 13.6]

6. Secondary Outcome: Time to Hepatic Progression (TTHP)
Description: Time to hepatic progression (TTHP) was defined as a period of time from the first on-study DEB-TACE till development of radiographic evidence of disease progression in the liver by mRECIST.
Time Frame: 1 year
Measure: Median (Full Range); unit: Months
Arm/Group | DEB-TACE
Number analyzed (Participants) | 17
Months | 5.9 [0.9 to 13.6]

7. Secondary Outcome: Progression Free Survival (PFS) Rate
Description: Progression free survival rate was defined as the number of patients who were alive and free from radiographic progression by mRECIST at pre-defined time periods.
  PFS rate was calculated at 3 months, 6 months, 12 months, and 24 months
Time Frame: 3 months, 6 months, 12 Months, and 24 months
Measure: Number; unit: participants
Arm/Group | DEB-TACE
Number analyzed (Participants) | 17
participants
  3 months | 14
  6 months | 10
  12 months | 6
  24 months | 4

8. Secondary Outcome: Proportion of Patients With Alpha-fetoprotein (AFP) Response With ≥ 50% Decline From Baseline
Description: This measure was defined as the number of patients with alpha-fetoprotein (AFP) response with ≥ 50% decline from baseline (in patients with baseline level ≥ 20) after DEB-TACE.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | DEB-TACE
Number analyzed (Participants) | 17
participants | 5

9. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Left ventricular ejection fraction (LVEF) was measured as percent contraction prior to the first DEB-TACE and 1 month following last planned DEB-TACE. Median LVEF and full range were reported.
Time Frame: Baseline, 1 month following last planned DEB-TACE
Measure: Median (Full Range); unit: percent contraction
Arm/Group | DEB-TACE
Number analyzed (Participants) | 17
percent contraction
  Baseline | 70 [66 to 81]
  1 month following last planned DEB-TACE | 68 [60 to 74]

10. Secondary Outcome: Median Area Under Curve (AUC)
Description: Area under curve for doxorubicin concentration in the serum over 7 days was measured by obtaining serum doxorubicin concentration samples at predose, 5 min, 20 min, 40 min, 60 min, 120 min, 6 hours, 24 hours, 7 days time points. A graph of serum doxorubicin concentration over time was then plotted for each of the 17 patients, and the area under the curve for each of the 17 patients was calculated.
  Pharmacokinetic sampling was performed only during each of the first planned DEB-TACE procedures.
Time Frame: 7 days
Measure: Median (Full Range); unit: ng/ml-hr
Arm/Group | DEB-TACE
Number analyzed (Participants) | 17
ng/ml-hr | 593 [175 to 2030]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | DEB-TACE
All-Cause Mortality (participants affected / at risk) | 12/17
Serious Adverse Events (participants affected / at risk) | 13/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DEB-TACE (N=17)
Hepatic failure (Gastrointestinal disorders) | 4
Ascites (Gastrointestinal disorders) | 1
Edema of legs (Musculoskeletal and connective tissue disorders) | 2
Hyperbilirubinemia (Gastrointestinal disorders) | 3
AST elevation (Gastrointestinal disorders) | 3
Hyponatremia (Renal and urinary disorders) | 4
Anemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DEB-TACE (N=17)
Anorexia (General disorders) | 6
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Fatigue (General disorders) | 8
Fever (General disorders) | 2
Hiccoughs (General disorders) | 1
Insomnia (General disorders) | 4
Nausea (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 6
ALT elevation (Gastrointestinal disorders) | 6
Creatinine elevation (Renal and urinary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT02147301/Prot_SAP_000.pdf